CLINICAL TRIAL: NCT03598114
Title: Program Sustainability Action Planning Training Project
Brief Title: Evaluating and Improving the Sustainability of State-level Tobacco Control Programs in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201801196; R01CA203844 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Program Sustainability; Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Sustainability Training (Experimental): * Selected publicly funded tobacco control programs receive the intervention in the form of custom training curricula designed to identify and enable sustainable tobacco control programming at a state-organizational level. Sustainability is assessed at t=12 months and 1=24 months to capture potential impact of the training and curricula.
  * The intervention group will receive a follow-up survey inviting them to evaluate the training and their progress on executing their sustainability plan. The intervention group will also receive a follow-up survey inviting them to evaluate the technical assistance they have received from the research team. Responses on neither follow-up survey impact participants standing in the study
  Interventions: Behavioral: Program Sustainability Action Planning Model and Training Curricula
- Control Condition (No Intervention): * In this condition, publicly funded tobacco control programs do not receive the designated program sustainability training and proceed with standard operations. Sustainability is assessed at t=12 months and t=24 months to compare against tobacco control programs receiving sustainability training
  * The control group will receive a follow-up survey inviting them to evaluate their progress on creating their sustainability plan. Responses on the follow-up survey do not impact participants' standing in the study

INTERVENTIONS:
Behavioral: Program Sustainability Action Planning Model and Training Curricula — The Program Sustainability Action Planning Model and Training Curricula's conceptual model is driven by the theory of change and incorporates aspects of Kolb's experiential learning theory to produce a six step process: defining the program, assessing the program, developing an action plan, executing the action plan, evaluating sustainability, and reassessing and modifying. The study team will deliver in-person, hand-on workshops incorporating each of these aspects of the conceptual model. Following the workshop, intervention states will partake in technical assistance activities with the study team to track progress and troubleshooting challenges.
  Arms: Program Sustainability Training

SUMMARY:
The purpose of this study is to empirically develop, test, and disseminate sustainability training to improve the institutionalization of evidence-based state tobacco control (TC) programs, and thus, tobacco-related health outcomes.

DETAILED DESCRIPTION:
This study defines program sustainability as the ability to maintain programming and its benefits over time.

The project builds upon the empirically-developed Program Sustainability Action Planning Model and Training Curricula. The training will incorporate experiential learning methods and includes: action planning workshops, development of action plans with measurable objectives to foster institutional changes, and technical assistance. The goal is to demonstrate change in sustainability outcomes in states who receive the Program Sustainability Action Planning Training compared to states that do not. After conclusion of the study, the sustainability training curriculum will be disseminated to all participating state TC programs. Additionally, the curriculum will be adapted for the use by any public health program in need of building sustainability capacity.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be non-institutionalized adults ages 18 and older.

Exclusion Criteria:

* Participants must be involved in their state's tobacco control program and must be selected by their state's Program Manager to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Luke, PhD, Study Chair — Center for Public Health Systems Science; Ross C Brownson, PhD, Study Chair — Prevention Research Center in St. Louis; Sarah Moreland-Russell, PhD, MPH, Principal Investigator — Prevention Research Center in St. Louis
Locations (1):
- Prevention Research Center in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gannon J, Moreland-Russell S. A qualitative study examining the impact of COVID-19 on capacity for sustainability of tobacco control programs. BMC Health Serv Res. 2024 Feb 16;24(1):215. doi: 10.1186/s12913-024-10633-9. PMID 38365656
- [Derived] Moreland-Russell S, Combs T, Gannon J, Jost E, Farah Saliba L, Prewitt K, Luke D, Brownson RC. Action planning for building public health program sustainability: results from a group-randomized trial. Implement Sci. 2024 Feb 2;19(1):9. doi: 10.1186/s13012-024-01340-4. PMID 38308331
- [Derived] Moreland-Russell S, Combs T, Gannon J, Jost E, Saliba LF, Prewitt K, Luke D, Brownson RC. Action Planning for Building Program Sustainability: Results from a Group-Randomized Trial. Res Sq [Preprint]. 2023 May 19:rs.3.rs-2783056. doi: 10.21203/rs.3.rs-2783056/v1. PMID 37292588
- [Derived] Moreland-Russell S, Jost E, Gannon J. A conceptual model for building program sustainability in public health settings: Learning from the implementation of the program sustainability action planning model and training curricula. Front Health Serv. 2023 Mar 29;3:1026484. doi: 10.3389/frhs.2023.1026484. eCollection 2023. PMID 37063373
- [Derived] Vitale R, Blaine T, Zofkie E, Moreland-Russell S, Combs T, Brownson RC, Luke DA. Developing an evidence-based program sustainability training curriculum: a group randomized, multi-phase approach. Implement Sci. 2018 Sep 26;13(1):126. doi: 10.1186/s13012-018-0819-5. PMID 30257695
- See also: This website provides a general project description. — https://prcstl.wustl.edu/items/plans-actions-and-capacity-to-sustain-tobacco-control-pact/
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine. — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 state tobacco-control programs were randomized to either the intervention group or the control group. Stakeholders from those state tobacco-control programs were consented and enrolled and the participant flow indicates the stakeholders that started and completed the trial.
Units Other Than Participants: State Tobacco Control Programs
Period: Overall Study
Arm/Group | Program Sustainability Training | Control Condition
Started | 127; 11 State Tobacco Control Programs | 128; 12 State Tobacco Control Programs
Completed | 124; 11 State Tobacco Control Programs | 89; 12 State Tobacco Control Programs
Not Completed | 3; 0 State Tobacco Control Programs | 39; 0 State Tobacco Control Programs
Not completed — Staff turnover/left the program | 3 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Program Sustainability Training | Control Condition | Total
Number analyzed (Participants) | 127 | 128 | 255
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 3 | 6 | 9
  30-39 years | 18 | 19 | 37
  40-49 years | 20 | 28 | 48
  50-59 years | 17 | 18 | 35
  60-69 years | 8 | 11 | 19
  70-79 years | 2 | 1 | 3
  Unknown or not reported age | 59 | 45 | 104
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 61 | 67 | 128
  Male | 14 | 19 | 33
  Unknown or not reported | 52 | 42 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 72 | 82 | 154
  Unknown or Not Reported | 54 | 44 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 7 | 5 | 12
  White | 57 | 74 | 131
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 55 | 45 | 100
Region of Enrollment [Number; unit: participants]
  United States | 127 | 128 | 255

OUTCOME MEASURES:

1. Primary Outcome: Change in Program Sustainability Assessment Tool (PSAT) Sustainability Scores
Description: The Program Sustainability Assessment Tool (PSAT) allows stakeholders to rate their programs on the extent to which they have processes and structures in place that will increase the likelihood of sustainability. The minimum score is 1 and the maximum score is 7. A higher score indicates greater program capacity for sustainability. Assessment results can be used to identify next steps in building program capacity for sustainability in order to position efforts for long term success.
Time Frame: 0 months,12 months, 24 months
Population: The results are the state's tobacco control program PSAT sustainability scores at each timepoint.
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- State 1 - Program Sustainability Training; State 4 - Program Sustainability Training; State 6 - Program Sustainability Training; State 8 - Program Sustainability Training; State 9 - Program Sustainability Training; State 11 - Program Sustainability Training; State 13 - Program Sustainability Training; State 15 - Program Sustainability Training; State 18 - Program Sustainability Training; State 19 - Program Sustainability Training; State 21 - Program Sustainability Training: * Selected publicly funded tobacco control programs receive the intervention in the form of custom training curricula designed to identify and enable sustainable tobacco control programming at a state-organizational level. Sustainability is assessed at t=12 months and 1=24 months to capture potential impact of the training and curricula.
  * The intervention group will receive a follow-up survey inviting them to evaluate the training and their progress on executing their sustainability plan. The intervention group will also receive a follow-up survey inviting them to evaluate the technical assistance they have received from the research team. Responses on neither follow-up survey impact participants standing in the study
- State 2 - Control Condition; State 3 - Control Condition; State 5 - Control Condition; State 7 - Control Condition; State 10 - Control Condition; State 12 - Control Condition; State 14 - Control Condition; State 16 - Control Condition; State 17 - Control Condition; State 20 - Control Condition; State 22 - Control Condition; State 23 - Control Condition: * In this condition, publicly funded tobacco control programs do not receive the designated program sustainability training and proceed with standard operations. Sustainability is assessed at t=12 months and t=24 months to compare against tobacco control programs receiving sustainability training
  * The control group will receive a follow-up survey inviting them to evaluate their progress on creating their sustainability plan. Responses on the follow-up survey do not impact participants' standing in the study
Arm/Group | State 1 - Program Sustainability Training | State 2 - Control Condition | State 3 - Control Condition | State 4 - Program Sustainability Training | State 5 - Control Condition | State 6 - Program Sustainability Training | State 7 - Control Condition | State 8 - Program Sustainability Training | State 9 - Program Sustainability Training | State 10 - Control Condition | State 11 - Program Sustainability Training | State 12 - Control Condition | State 13 - Program Sustainability Training | State 14 - Control Condition | State 15 - Program Sustainability Training | State 16 - Control Condition | State 17 - Control Condition | State 18 - Program Sustainability Training | State 19 - Program Sustainability Training | State 20 - Control Condition | State 21 - Program Sustainability Training | State 22 - Control Condition | State 23 - Control Condition
Number analyzed (Participants) | 31 | 22 | 9 | 24 | 14 | 22 | 12 | 20 | 20 | 31 | 31 | 14 | 25 | 31 | 40 | 24 | 18 | 19 | 11 | 25 | 17 | 28 | 11
score on a scale
  0 months: number analyzed (Participants) | 13 | 7 | 7 | 10 | 7 | 9 | 9 | 12 | 9 | 15 | 14 | 6 | 7 | 11 | 12 | 11 | 9 | 10 | 6 | 12 | 8 | 11 | 5
  0 months | 4.9 (0.7) | 5.1 (0.4) | 3.8 (0.5) | 4.2 (0.5) | 5.1 (0.8) | 5.0 (0.5) | 5.3 (0.6) | 5.2 (0.5) | 4.4 (0.7) | 4.5 (0.5) | 4.5 (0.4) | 3.8 (1.1) | 4.7 (0.5) | 5.4 (0.5) | 4.3 (0.4) | 4.5 (0.6) | 4.4 (0.6) | 4.0 (0.4) | 4.3 (0.6) | 4.2 (0.6) | 4.1 (0.5) | 4.2 (0.4) | 2.9 (0.6)
  12 months: number analyzed (Participants) | 10 | 5 | 1 | 8 | 6 | 7 | 2 | 4 | 5 | 8 | 8 | 4 | 10 | 11 | 8 | 5 | 5 | 4 | 4 | 5 | 5 | 9 | 3
  12 months | 5.2 (0.6) | 5.4 (0.6) | 5.0 (0.8) | 4.0 (0.4) | 5.1 (0.8) | 5.0 (0.5) | 6.0 (0.5) | 5.7 (0.2) | 3.5 (0.7) | 4.3 (0.4) | 4.3 (0.2) | 3.4 (0.6) | 4.9 (0.5) | 4.9 (0.4) | 3.6 (0.6) | 5.5 (0.4) | 4.9 (0.5) | 3.9 (0.4) | 4.6 (0.3) | 4.5 (0.9) | 4.5 (0.8) | 4.4 (0.4) | 2.8 (0.5)
  24 months: number analyzed (Participants) | 8 | 10 | 1 | 6 | 1 | 6 | 1 | 4 | 6 | 8 | 9 | 4 | 8 | 9 | 20 | 8 | 4 | 5 | 1 | 8 | 4 | 8 | 3
  24 months | 5.4 (0.7) | 5.2 (0.4) | 4.5 (1.3) | 4.2 (0.3) | 5.8 (1.0) | 5.3 (0.5) | 5.5 (0.8) | 5.7 (0.5) | 3.7 (0.5) | 4.5 (0.7) | 4.7 (0.4) | 3.7 (0.6) | 5.2 (0.5) | 5.0 (0.2) | 4.5 (0.3) | 5.0 (0.5) | 4.7 (0.5) | 4.0 (0.5) | 5.7 (0.7) | 4.1 (0.7) | 4.0 (0.8) | 4.6 (0.3) | 3.5 (0.7)

2. Secondary Outcome: Number of State Tobacco Control Programs Present in Law, Regulation, or Rule
Description: -This measure is defined as whether a state's tobacco control program is established or continued through state statute or regulation and/or if the program is stated in organizational doctrine as a permanent component of the auspice organization. This is a direct measure of formal institutionalization of tobacco control programs and will be measured as a simple binary quantity, zero (0) for "not present in law, regulation, or rule" and one (1) for "present in law, regulation, or rule."
Time Frame: 0 months, 12 months, 24 months
Population: The data for this outcome measure was gathered at a state level and not at the stakeholder level.
Measure: Count of Units; unit: State Tobacco Control Programs
Units Other Than Participants: State Tobacco Control Programs
Arm/Group | State 1 - Program Sustainability Training | State 2 - Control Condition | State 3 - Control Condition | State 4 - Program Sustainability Training | State 5 - Control Condition | State 6 - Program Sustainability Training | State 7 - Control Condition | State 8 - Program Sustainability Training | State 9 - Program Sustainability Training | State 10 - Control Condition | State 11 - Program Sustainability Training | State 12 - Control Condition | State 13 - Program Sustainability Training | State 14 - Control Condition | State 15 - Program Sustainability Training | State 16 - Control Condition | State 17 - Control Condition | State 18 - Program Sustainability Training | State 19 - Program Sustainability Training | State 20 - Control Condition | State 21 - Program Sustainability Training | State 22 - Control Condition | State 23 - Control Condition
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Number analyzed (State Tobacco Control Programs) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
State Tobacco Control Programs
  0 months | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  12 months | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  24 months | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0

3. Secondary Outcome: State Tobacco Control Program is Included as Part of Regular Budget
Description: Defined as whether a state's tobacco control program is a regular (annual, quarterly, or otherwise) item of the budget of its auspice organization. It directly indicated formal institutionalization and will take one of two possible values, zero (0) for "not included in budget" and one (1) for "included in budget."
Time Frame: 0 months, 12 months, 24 months
Population: The data for this outcome measure was gathered at a state level and not at the stakeholder level. The 12 month data time point for state 23 is missing.
Measure: Count of Units; unit: State Tobacco Control Programs
Units Other Than Participants: State Tobacco Control Programs
Arm/Group | State 1 - Program Sustainability Training | State 2 - Control Condition | State 3 - Control Condition | State 4 - Program Sustainability Training | State 5 - Control Condition | State 6 - Program Sustainability Training | State 7 - Control Condition | State 8 - Program Sustainability Training | State 9 - Program Sustainability Training | State 10 - Control Condition | State 11 - Program Sustainability Training | State 12 - Control Condition | State 13 - Program Sustainability Training | State 14 - Control Condition | State 15 - Program Sustainability Training | State 16 - Control Condition | State 17 - Control Condition | State 18 - Program Sustainability Training | State 19 - Program Sustainability Training | State 20 - Control Condition | State 21 - Program Sustainability Training | State 22 - Control Condition | State 23 - Control Condition
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Number analyzed (State Tobacco Control Programs) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
State Tobacco Control Programs
  0 months | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  12 months: number analyzed (State Tobacco Control Programs) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0
  12 months | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 |
  24 months | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1

4. Secondary Outcome: Change in Percentage of Organizational Budget Allotted to Tobacco Control Program
Description: Defined as the percentage of the state health department budget garnered by its tobacco control program. The measure will be continuous and theoretically range from 0% (no funding) to 100% (entire health department budget). This quantity measures institutionalization of a program both individually and relative to other state health programs.
Time Frame: 0 months, 12 months, 24 months
Population: The data for this outcome measure was gathered at a state level and not at the stakeholder level.
Measure: Number; unit: percentage of health department budget
Units Other Than Participants: State Tobacco Control Programs
Arm/Group | State 1 - Program Sustainability Training | State 2 - Control Condition | State 3 - Control Condition | State 4 - Program Sustainability Training | State 5 - Control Condition | State 6 - Program Sustainability Training | State 7 - Control Condition | State 8 - Program Sustainability Training | State 9 - Program Sustainability Training | State 10 - Control Condition | State 11 - Program Sustainability Training | State 12 - Control Condition | State 13 - Program Sustainability Training | State 14 - Control Condition | State 15 - Program Sustainability Training | State 16 - Control Condition | State 17 - Control Condition | State 18 - Program Sustainability Training | State 19 - Program Sustainability Training | State 20 - Control Condition | State 21 - Program Sustainability Training | State 22 - Control Condition | State 23 - Control Condition
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Number analyzed (State Tobacco Control Programs) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
percentage of health department budget
  0 months | 31.80 | 12.30 | 0.80 | 1.70 | 2.50 | 3.90 | 6.30 | 18.10 | 3.70 | 9.00 | 5.30 | 16.20 | 11.50 | 10.00 | 2.40 | 4.70 | 3.30 | 7.00 | 2.60 | 5.60 | 3.10 | 7.60 | 3.90
  12 months | 13.10 | 22.30 | 5.10 | 3.40 | 8.50 | 20.40 | 18.20 | 17.00 | 4.90 | 7.40 | 13.30 | 22.00 | 10.90 | 12.40 | 6.60 | 4.50 | 3.70 | 6.50 | 2.60 | 5.50 | 3.00 | 7.70 | 3.50
  24 months | 12.10 | 19.80 | 0.90 | 4.00 | 7.90 | 13.20 | 13.60 | 16.50 | 4.80 | 7.10 | 10.80 | 19.00 | 11.20 | 10.20 | 6.80 | 4.30 | 4.20 | 6.30 | 2.70 | 4.20 | 5.20 | 7.50 | 4.00

5. Secondary Outcome: Change in Percentage of CDC-recommended Tobacco Control Funding Level Actually Spent
Description: Defined as the amount of program funding as a percentage of the amount recommended by the CDC. This quantity measures institutionalization of a program relative to an objective level of funding computed uniformly from state characteristics by the CDC. The measure ranges from 0% (no funding) to over 100% (above CDC-recommended level).
Time Frame: 0 months, 12 months, 24 months
Population: The data for this outcome measure was gathered at a state level and not at the stakeholder level.
Measure: Number; unit: % of CDC-recommended funding spent
Units Other Than Participants: State Tobacco Control Programs
Arm/Group | State 1 - Program Sustainability Training | State 2 - Control Condition | State 3 - Control Condition | State 4 - Program Sustainability Training | State 5 - Control Condition | State 6 - Program Sustainability Training | State 7 - Control Condition | State 8 - Program Sustainability Training | State 9 - Program Sustainability Training | State 10 - Control Condition | State 11 - Program Sustainability Training | State 12 - Control Condition | State 13 - Program Sustainability Training | State 14 - Control Condition | State 15 - Program Sustainability Training | State 16 - Control Condition | State 17 - Control Condition | State 18 - Program Sustainability Training | State 19 - Program Sustainability Training | State 20 - Control Condition | State 21 - Program Sustainability Training | State 22 - Control Condition | State 23 - Control Condition
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Number analyzed (State Tobacco Control Programs) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
% of CDC-recommended funding spent
  0 months | 31.93 | 102.22 | 3.43 | 8.54 | 20.92 | 45.0 | 42.99 | 36.22 | 8.90 | 13.14 | 51.27 | 58.89 | 43.10 | 23.70 | 3.53 | 10.21 | 8.27 | 11.02 | 4.50 | 19.20 | 7.57 | 12.11 | 7.10
  12 months | 28.20 | 102.20 | 10.20 | 6.90 | 20.90 | 58.50 | 43.00 | 36.70 | 9.0 | 14.0 | 36.20 | 53.50 | 41.90 | 28.50 | 10.50 | 11.00 | 8.30 | 11.20 | 4.70 | 19.30 | 7.60 | 13.20 | 6.70
  24 months | 28.20 | 98.10 | 2.0 | 8.40 | 21.10 | 43.40 | 32.40 | 37.60 | 8.90 | 13.90 | 30.70 | 45.70 | 42.50 | 23.20 | 10.50 | 10.50 | 9.00 | 10.60 | 4.70 | 16.00 | 13.20 | 12.90 | 7.40

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events, and adverse events were collected from the start of trial through 24 month follow-up.
Arm/Group | Program Sustainability Training | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/128
Other Adverse Events (participants affected / at risk) | 0/127 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03598114/Prot_SAP_ICF_000.pdf